CLINICAL TRIAL: NCT06246019
Title: The Clinical Impact of the Novel Alzheimer's Blood-based Biomarkers: the PLASMAR Study
Brief Title: The Clinical Impact of the Novel Alzheimer's Blood-based Biomarkers
Acronym: PLASMAR
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospital del Mar Research Institute (IMIM) (Other)
Responsible Party: Principal Investigator, Marc Suarez-Calvet, Head of the Fluid Biomarkers and Translational Neurology Research Group, Hospital del Mar Research Institute (IMIM)
Other Study IDs: 15225
Record Dates: First submitted 2024-01-23; First posted 2024-02-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer Disease; Cognitive Impairment; Dementia; Neurodegenerative Diseases; Frontotemporal Dementia; Lewy Body Disease; Vascular Dementia
Keywords: Blood-biomarkers; Alzheimer Disease; Diagnosis; Dementia; Cognitive impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Neurodegenerative Diseases; Frontotemporal Dementia; Lewy Body Disease; Dementia, Vascular; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid samples, serum and plasma samples will be processed and stored in the BIODEGMAR collection at the facilities of the Hospital del Mar Research Institute (IMIM). The sample collection of the present study has been registered in the National Registry of Biobanks, Instituto de Salud Carlos III (ISCIII), code: 0005744.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Blood-based biomarkers Arm: The results of the blood-based biomarkers will be communicated to the managing neurologist at visit 1 (at 3 months from baseline visit).
  Interventions: Diagnostic Test: Early adoption of blood-based biomarkers for Alzheimer's disease
- Late Blood-based biomarkers Arm: The results of the blood-based biomarkers will be communicated to the managing neurologist at visit 2 (at 9 months from baseline visit).
  Interventions: Diagnostic Test: Early adoption of blood-based biomarkers for Alzheimer's disease

INTERVENTIONS:
Diagnostic Test: Early adoption of blood-based biomarkers for Alzheimer's disease — A blood test will be performed to obtain plasma measures of Amyloid-β (Aβ) 42/40, phosphorylated tau (p-tau) 181, p-tau217, p-tau231 and Glial fibrillary acidic protein (GFAP) and Neurofilament light chain (NfL) and results will be disclosure to the early and late arms at different time points.

SUMMARY:
The goal of this observational study is to determine whether the early adoption of blood-based biomarkers for Alzheimer's disease is associated with an impact on etiological diagnosis, patient's management, emotional impact, patient's preferences and cost-effectiveness in patients presenting with cognitive complaints in a Cognitive Disorders Unit from a public hospital.

The main questions it aims to answer are:

1. Does the early adoption of blood-based biomarkers in clinical practice enable an earlier etiologic diagnosis with high confidence compared to the late adoption of blood-based biomarkers in the patients with cognitive complaints that are admitted in a Cognitive Disorders Unit?
2. Is the early adoption of blood-based biomarkers in clinical practice associated with changes in clinical management compared to their late adoption?
3. Is the early adoption of blood-based biomarkers in clinical practice associated with a lower emotional impact in the patients and their study partners/caregivers compared to their late adoption?
4. Are blood-based biomarkers better tolerated than other tests and preferred by patients for the diagnostic work-up?
5. Does blood-based biomarkers have an impact in the cost of the diagnostic workup and clinical management of the patients that are admitted in a Cognitive Disorders Unit?

Participants will be asked to:

* Perform a blood extraction for blood-based biomarkers analysis at the beginning of the study.
* Complete specific scales in each visit.

Researchers will compare the group in which blood biomarkers are delivered at 3 months with the group in which they are delivered at 9 months to assess whether early adoption of blood-based biomarkers is associated with an impact on etiological diagnosis, patient's management, emotional impact, patient's preferences and cost-effectiveness in a specialized memory unit.

DETAILED DESCRIPTION:
Blood-based biomarkers that accurately detect Alzheimer's disease (AD) and neurodegeneration now offer a realistic, cost-effective and non-invasive assessment that will aid the diagnostic process in patients presenting with cognitive clinical manifestations. Plasma measures of Amyloid-β (Aβ) 42/40, phosphorylated tau (p-tau) 181, p-tau217, p-tau231 and Glial fibrillary acidic protein (GFAP) have shown high diagnostic accuracy to detect AD, while plasma Neurofilament light chain (NfL) indicates neuronal injury. Despite these promising results, there is still no clear real-word evidence of their clinical applications. Here, the PLASMAR project aims to determine whether blood-based biomarkers have an impact on the clinical management of patients presenting with cognitive complaints in a Cognitive Disorders Unit from a public hospital, which provides care to a heterogeneous population. The project is divided into two specific objectives. First, the investigators will determine, in a research cohort, which blood biomarker or biomarkers' combination have the highest accuracy to detect AD. Second, a prospective clinical cohort of consecutive patients coming to the memory unit will be recruited. The investigators will assess whether early adoption of blood-based biomarkers is associated with an impact on etiological diagnosis, patient's management, emotional impact, patient's preferences and cost-effectiveness in a specialized memory unit. Answering the question of whether blood-based biomarkers have a clinical impact in the real-world scenario of a memory unit, the PLASMAR project is crucial for the healthcare system and can guide the developing of guidelines and protocols on the use of blood-based biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 and ≤85 years old of any sex, gender, race or ethnicity.
* Individuals interested in participating in the study who understand the procedures that will be performed.
* The patient must have a complaint (reported by the patient or by a study partner/caregiver) of cognitive or behavioral impairment.
* The patient must satisfy the clinical diagnostic criteria for subjective cognitive decline, mild cognitive impairment, or mild dementia (defined as a Global deterioration scale score equal to 4), and a neurodegenerative disease such as AD is considered in the differential diagnosis.
* Agreement to undergo all the study procedures, complete all clinical visits according to protocol and capacity to give informed consent.
* The patient has undergone (maximum 12 months ago) or will undergo a dementia blood workup and MRI and/or CT scan before V1.
* In dementia patients, a study partner must be available for the duration of the protocol.

Exclusion Criteria:

* Any significant systemic illness or unstable medical condition that could make it difficult to comply with the protocol.
* Medical contraindications for any of the study procedures.
* Available AD's cerebrospinal fluid biomarkers levels or amyloid-PET at screening.
* The patient comes to the Memory Unit for reasons other than cognitive or behavioral impairment.
* Patients in which an etiological diagnosis is already made.
* The patient is currently participating or has participated in a clinical trial with an investigational pharmaceutical product.
* Women who are pregnant, planning to become pregnant, or lactating.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PLASMAR is prospective, unicentric, unblinded and randomized controlled study with blinded outcome ascertainment. Two hundred new patients will be consecutively recruited. All consecutive new patients who are visited for the first time to the outpatients' Memory Clinic at the Neurology Service (Hospital del Mar, Barcelona, Spain) will be considered for the study. Each patient will name a study partner to participate in this study, who will be considered for the study as well. In case the patient is diagnosed with dementia, a caregiver will be considered.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Etiological diagnosis | 9 months
  The proportion of patients for whom an etiologic diagnosis is reached with very high confidence (≥90%) in each group at 3 and 9 months.
Suspicion of neurodegenerative disease | 9 months
  The proportion of patients for whom a suspicion of neurodegenerative disease is reached as etiology with very high confidence (≥90%) in each group at 3 and 9 months.

SECONDARY OUTCOMES:
Number of tests for etiological diagnosis | 9 months
  The number of tests necessary to reach an etiological diagnosis with very high confidence (≥90%) in each group at 3 and 9 months.
Number of tests for a suspicion of neurodegenerative disease | 9 months
  The number of tests to reach a suspicion of neurodegenerative disease as etiology with very high confidence (≥90%) in each group at 3 and 9 months.
Neurologist diagnoses over time | 9 months
  Changes in the neurologist's etiologic diagnosis in each group during the time of the study.
Neurologist confidence in the etiological diagnosis, which is is collected through the PLASMAR questionnaire at each visit. | 9 months
  Changes in the neurologist's estimate of the likelihood that the patient's symptoms are due to AD in each group during the time of the study.
Neurologist confidence in the suspicion of neurodegenerative disease, which is is collected through the PLASMAR questionnaire at each visit. | 9 months
  Changes in the neurologist's estimate of the likelihood that the patient's symptoms are due to a neurodegenerative disease as etiology in each group during the time of the study.

OTHER OUTCOMES:
Number of patients whose clinical management in the Cognitive Disorders Unit changes | 9 months
  Changes in the prescription or withdrawal of disease-specific pharmacologic treatments (cholinesterase inhibitors, Memantine) and other pharmacologic or non-pharmacological interventions in addition to the number of patients who are discharged from the Cognitive Disorders Unit during the time of the study.
Emotional impact of blood-based biomarkers on patient and study partner/caregiver | 9 months
  Changes in Hospital Anxiety and Depression Scale (HADS; score: 0-42, with higher scores indicating higher anxiety or depression) and The Perceived Stress Scale (PSS; score: 0-40, with higher scores indicating higher perceived stress) during the time of the study.
Impact of blood-based biomarkers on patient's quality of life | 9 months
  Changes in the 5-level European Quality of Life-5 Dimensions scale (EQ-5D-5L; score: 5-25, with higher scores indicating worse severity index) during the time of the study.
Patient's tolerance to biomarkers tests and their preferences in how they want to be diagnosed | 9 months
  Tolerance score for each of the tests performed as part of clinical practice during the time of the study.
Relative cost savings from the Implementation of blood-based biomarkers in the Cognitive Disorders Unit. | 9 months
  The cost of the diagnostic work-up to achieve an etiologic diagnosis with very high confidence (≥90%) and the cost savings in resources (arising from pharmacological or non-pharmacological interventions, as well as discharges) will be combined to determine the relative cost of implementing blood-based biomarkers compared to their non-implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Suárez-Calvet, MD PhD, Principal Investigator — Hospital del Mar Research Insititute (IMIM); Albert Puig-Pijoan, MD, Principal Investigator — Hospital del Mar Research Insititute (IMIM)
Locations (1):
- Hospital del Mar, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Altomare D, Barkhof F, Caprioglio C, Collij LE, Scheltens P, Lopes Alves I, Bouwman F, Berkhof J, van Maurik IS, Garibotto V, Moro C, Delrieu J, Payoux P, Saint-Aubert L, Hitzel A, Molinuevo JL, Grau-Rivera O, Gispert JD, Drzezga A, Jessen F, Zeyen P, Nordberg A, Savitcheva I, Jelic V, Walker Z, Edison P, Demonet JF, Gismondi R, Farrar G, Stephens AW, Frisoni GB; Amyloid Imaging to Prevent Alzheimer's Disease (AMYPAD) Consortium. Clinical Effect of Early vs Late Amyloid Positron Emission Tomography in Memory Clinic Patients: The AMYPAD-DPMS Randomized Clinical Trial. JAMA Neurol. 2023 Jun 1;80(6):548-557. doi: 10.1001/jamaneurol.2023.0997. PMID 37155177
- [Background] Grothe MJ, Moscoso A, Ashton NJ, Karikari TK, Lantero-Rodriguez J, Snellman A, Zetterberg H, Blennow K, Scholl M; Alzheimer's Disease Neuroimaging Initiative. Associations of Fully Automated CSF and Novel Plasma Biomarkers With Alzheimer Disease Neuropathology at Autopsy. Neurology. 2021 Sep 20;97(12):e1229-e1242. doi: 10.1212/WNL.0000000000012513. PMID 34266917
- [Background] Janelidze S, Mattsson N, Palmqvist S, Smith R, Beach TG, Serrano GE, Chai X, Proctor NK, Eichenlaub U, Zetterberg H, Blennow K, Reiman EM, Stomrud E, Dage JL, Hansson O. Plasma P-tau181 in Alzheimer's disease: relationship to other biomarkers, differential diagnosis, neuropathology and longitudinal progression to Alzheimer's dementia. Nat Med. 2020 Mar;26(3):379-386. doi: 10.1038/s41591-020-0755-1. Epub 2020 Mar 2. PMID 32123385
- [Background] Karikari TK, Pascoal TA, Ashton NJ, Janelidze S, Benedet AL, Rodriguez JL, Chamoun M, Savard M, Kang MS, Therriault J, Scholl M, Massarweh G, Soucy JP, Hoglund K, Brinkmalm G, Mattsson N, Palmqvist S, Gauthier S, Stomrud E, Zetterberg H, Hansson O, Rosa-Neto P, Blennow K. Blood phosphorylated tau 181 as a biomarker for Alzheimer's disease: a diagnostic performance and prediction modelling study using data from four prospective cohorts. Lancet Neurol. 2020 May;19(5):422-433. doi: 10.1016/S1474-4422(20)30071-5. PMID 32333900
- [Background] Simren J, Andreasson U, Gobom J, Suarez Calvet M, Borroni B, Gillberg C, Nyberg L, Ghidoni R, Fernell E, Johnson M, Depypere H, Hansson C, Jonsdottir IH, Zetterberg H, Blennow K. Establishment of reference values for plasma neurofilament light based on healthy individuals aged 5-90 years. Brain Commun. 2022 Jul 4;4(4):fcac174. doi: 10.1093/braincomms/fcac174. eCollection 2022. PMID 35865350
- [Background] Suarez-Calvet M, Karikari TK, Ashton NJ, Lantero Rodriguez J, Mila-Aloma M, Gispert JD, Salvado G, Minguillon C, Fauria K, Shekari M, Grau-Rivera O, Arenaza-Urquijo EM, Sala-Vila A, Sanchez-Benavides G, Gonzalez-de-Echavarri JM, Kollmorgen G, Stoops E, Vanmechelen E, Zetterberg H, Blennow K, Molinuevo JL; ALFA Study. Novel tau biomarkers phosphorylated at T181, T217 or T231 rise in the initial stages of the preclinical Alzheimer's continuum when only subtle changes in Abeta pathology are detected. EMBO Mol Med. 2020 Dec 7;12(12):e12921. doi: 10.15252/emmm.202012921. Epub 2020 Nov 10. PMID 33169916
- [Background] Thijssen EH, La Joie R, Strom A, Fonseca C, Iaccarino L, Wolf A, Spina S, Allen IE, Cobigo Y, Heuer H, VandeVrede L, Proctor NK, Lago AL, Baker S, Sivasankaran R, Kieloch A, Kinhikar A, Yu L, Valentin MA, Jeromin A, Zetterberg H, Hansson O, Mattsson-Carlgren N, Graham D, Blennow K, Kramer JH, Grinberg LT, Seeley WW, Rosen H, Boeve BF, Miller BL, Teunissen CE, Rabinovici GD, Rojas JC, Dage JL, Boxer AL; Advancing Research and Treatment for Frontotemporal Lobar Degeneration investigators. Plasma phosphorylated tau 217 and phosphorylated tau 181 as biomarkers in Alzheimer's disease and frontotemporal lobar degeneration: a retrospective diagnostic performance study. Lancet Neurol. 2021 Sep;20(9):739-752. doi: 10.1016/S1474-4422(21)00214-3. PMID 34418401
- See also: Fluid Biomarkers and Translational Neurology group — https://www.imim.cat/programesrecerca/neurociencies/en_biomarcadors_fluids_neurologia.html